CLINICAL TRIAL: NCT04111185
Title: Blood Volume Analysis - Guided Heart Failure Management
Brief Title: Daxor - Blood Volume Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00102851
Record Dates: First submitted 2019-09-23; First posted 2019-10-01 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Receive Blood Volume Analysis Guided Treatment (Experimental): The health care team will be provided with BVA results and may use the information to make decisions regarding the participant's treatment.
  Interventions: Device: Receive Blood Volume Analysis Guided Treatment
- Receive Standard of Care Treatment (No Intervention): The health care team will not be provided with the BVA results. The participant will receive the same treatment they would have received if they weren't in the study.

INTERVENTIONS:
Device: Receive Blood Volume Analysis Guided Treatment — The health care team will be given the results of the blood volume analysis along with guidance on how to provide treatment based on the analysis
  Other Names: Daxor BVA-100
  Arms: Receive Blood Volume Analysis Guided Treatment

SUMMARY:
The purpose of this study is to better understand blood volume status and whether knowledge of it can change and improve heart failure care.

DETAILED DESCRIPTION:
The purpose of this study is to better understand measurements of various parameters of congestion, the most significant of which is blood volume analysis. Blood volume analysis (BVA) measures how much blood is in the investigator's arteries and veins and is performed by using an IV and injecting a small amount of a radioactive material (I 131-labeled albumin). The study also involves blood tests, urine tests, blood pressure monitoring, an ultrasound, and measurement of lung fluid volume (by way of a vest). There will also be a 30-day follow-up phone call to assess symptoms and discuss any changes in medication.

ELIGIBILITY:
Inclusion Criteria:

- Admission for acute decompensated heart failure to the cardiology service at Duke Hospital, Durham, North Carolina

Exclusion Criteria:

* Age < 18 years
* Ongoing pregnancy
* Recent acute MI or hemodynamic instability: Acute MI (STEMI or Type I NSTEMI) within 7 days
* Post heart transplantation or ongoing mechanical circulatory support
* Progressive cardiogenic shock
* Patients with Ventricular Assist Devices
* End stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Michael Felker, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Receive Blood Volume Analysis Guided Treatment: The health care team will be provided with BVA (blood volume analysis) results and may use the information to make decisions regarding the participant's treatment.
  Receive Blood Volume Analysis Guided Treatment: The health care team will be given the results of the blood volume analysis along with guidance on how to provide treatment based on the analysis
Period: Overall Study
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Started | 17 | 14
Completed | 17 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (32) | 60 (30) | 61 (31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Whole Blood Volume
Time Frame: Baseline, and upon discharge (up to day 18)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Number analyzed (Participants) | 17 | 14
mL | -1253 (2157) | -784 (981)
Statistical Analysis 1: Comparison: Receive Blood Volume Analysis Guided Treatment vs Receive Standard of Care Treatment; Test type: Other; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Change in Congestion Metrics as Measured With a Clinical Congestion Score (Pulmonary Edema, Jugular Venous Pressure, Lower Extremity Edema and PND)
Description: Comparison of baseline to follow up times
Time Frame: Baseline, day 1, day 2, day 3 and discharge (up to day 18)
Population: Data not collected.
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Mean NTpro-BNP Concentration (in pg/mL)
Time Frame: Baseline, day 1, day 2, day 3 and discharge (up to day 18); reported as change from baseline to discharge
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Number analyzed (Participants) | 17 | 14
pg/mL | -853 (3154) | -4849 (6770)

4. Secondary Outcome: Change in Weight (in kg)
Time Frame: Baseline, day 1, day 2, day 3 and discharge (up to day 18); reported as change from baseline to discharge
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Number analyzed (Participants) | 17 | 14
kg | -6.4 (5.4) | -10.1 (10.6)

5. Secondary Outcome: Change in Renal Function as Measured by Creatinine (mg/dL)
Time Frame: Baseline, day 1, day 2, day 3 and discharge (up to day 18); reported as change from baseline to discharge
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Number analyzed (Participants) | 17 | 14
mg/dL | 0.1 (0.3) | 0.2 (0.3)

6. Secondary Outcome: Change in Renal Function as Measured by Blood Urea Nitrogen (mg/dL)
Description: Comparison of baseline to follow up times
Time Frame: Baseline, day 1, day 2, day 3 and discharge (up to day 18)
Population: Data not collected.
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Renal Function as Measured by an Estimated Glomerular Filtration Rate (mL/Min/ 1.73m2)
Description: Comparison of baseline to follow up times
Time Frame: Baseline, day 1, day 2, day 3 and discharge (up to day 18)
Population: Data not collected.
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Pulmonary Congestion as Measured Using Non-invasive Diagnostic Technology Such as the ReDS Vest (Radiofrequency) or Bio-impedance Based Technologies (Unitless Values)
Description: Comparison of baseline to follow up times
Time Frame: Baseline, day 1, day 2, day 3 and discharge (up to day 18)
Population: Data not collected.
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 18 days
Arm/Group | Receive Blood Volume Analysis Guided Treatment | Receive Standard of Care Treatment
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT04111185/Prot_SAP_000.pdf